CLINICAL TRIAL: NCT06522451
Title: Effects of Conventional Physical Therapy With and Without Cuevas Medek Exercises on Gross Motor Function in Children With Motor Developmental Delay
Brief Title: Effects of Conventional Physical Therapy With and Without Cuevas Medek Exercises in Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/07106
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Motor Delay
Keywords: Cuevas Medek exercises; developmental delay
MeSH Terms: conditions — Psychomotor Disorders; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: It will be Randomized control trial in which non probability convenient sampling will be used. Two groups of age 12-42 months will be formed in which participants will be randomly divided. Group A will only receive conventional physical therapy and group B will receive conventional physical therapy with cuevas medek exercises
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy (Active Comparator): This group receives conventional physical therapy
  Interventions: Other: conventional physical therapy
- Conventional physical therapy with cuevas medek exercises (Experimental): This group receives conventional physical therapy along with cuevas medek exercises
  Interventions: Other: Conventional physical therapy along with cuevas medek exercises

INTERVENTIONS:
Other: conventional physical therapy — Only conventional physical therapy (CPT) will be administered to this group. These regular workouts will include dynamic and static stretching, walking-specific functional exercises, passive mobilizations for pain-free mobility, balance modulation, and gait training. At baseline, the functional state of both groups will be evaluated. Treatment sessions will run for a total of 12 weeks, five days a week, for 45 minutes each. They will consist of four to six repeated exercises, six times on average, and use BSID-4 once the trial is over.
  Arms: Conventional Physical Therapy
Other: Conventional physical therapy along with cuevas medek exercises — In addition to regular physical therapy, this group will get Cuevas Medak exercises including head and trunk control (by stabilizing limb) and standing to sitting transition. For a duration of 12 weeks, five days a week, and 45 minutes, each session will be held. At the baseline, the functional state of both groups will be evaluated.
  Arms: Conventional physical therapy with cuevas medek exercises

SUMMARY:
There are several etiologies for developmental delay (DD). One of the main causes of developmental delay is cerebral palsy (CP), which has a variety of clinical characteristics brought on by damage to the developing brain. Children with developmental delays frequently have difficulties with feeling, perception, cognition, communication, musculoskeletal disorders, and movement and posture. A child's developmental delay could be avoided and motor milestones could be reached with the help of a CME-based intervention. In order to lessen or prevent developmental motor delay, CME-based intervention may be taken into consideration as a research issue and as an option for either intensive or conventional therapy.

A randomized control trial will be used for this. The Sehat Medical Complex in Lahore's physiotherapy department would be the source of the data collection. This study includes children of any gender between the ages of 12 and 42 months. Babies with motor developmental delays are diagnosed and their treatment plans are developed using the Bayley Scales of Infants and Toddlers IV (BSID-4). Conventional physical treatment, including dynamic/static stretches, functional exercises, passive mobilizations, balance modulation, and gait training, was administered to group A. At baseline, the functional state of both groups will be evaluated. Treatment sessions will run for a total of 12 weeks, five days a week, for 45 minutes each. They will consist of four to six repeated exercises, six times on average, and will continue to use BSID-4 after the study is finished. Group B includes Cuevas Medak exercises like transition and head and trunk control (by stabilizing limb) and sitting-to-standing transition are recommended. For a duration of 12 weeks, five days a week, and 45 minutes, each session will be held. At baseline, the functional state of both groups will be evaluated. then once the sessions are over, more data will be gathered using BSID-4. This research will help determine the efficacy of CME therapy in addition to traditional physical therapy.

DETAILED DESCRIPTION:
Group A: Control Group: The only form of physical therapy (CPT) given to this group will be conventional CPT. These regular workouts will include dynamic and static stretching, walking-specific functional exercises, passive mobilizations for pain-free mobility, balance modulation, and gait training. At baseline, the functional state of both groups will be evaluated. Treatment sessions will run for a total of 12 weeks, five days a week, for 45 minutes each. They will consist of four to six repeated exercises, six times on average, and use BSID-4 once the trial is over.

Group B: Experimental Group: In addition to regular physical therapy, this group will also get Cuevas Medak exercises, such as head and trunk control (by stabilizing limb) and standing to sitting transition. For a duration of 12 weeks, five days a week, and 45 minutes, each session will be held. At baseline, the functional state of both groups will be evaluated. then once the sessions are over, more data will be gathered using BSID-4.

ELIGIBILITY:
Inclusion Criteria:

* Children with motor developmental delay will only be included, and it will be ruled out by using Portage's Guide.
* Age between 12 and 42 months.
* Both genders

Exclusion Criteria:

* Individuals who suffer from particular neurological impairments, such as hydrocephalus, or who have related conditions.
* Patients with systemic disorders, infectious diseases, or vision impairment will not be accepted.
* Spinal surgery history

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Infant and toddler Development IV | 12 weeks
  The Bayley scales of infants and toddlers IV (BSID-4) is an individually administered instrument that evaluates the developmental functioning of infants and young children between the ages of one and forty-two months. There are two ways to administer the BSID-4: the Social-Emotional and Adaptive Behavior scales, which is a questionnaire that parents or caregivers complete, and the Cognitive, Language, and Motor scales, which are administered by a qualified professional and scored through observation and direct interaction with the child. To obtain qualitative information about motor skills (e.g., attends to the examiner on camera, shifts attention when name is called, babbles, reaches and groups objects), the BSID-4 contains 56 items in the gross motor domain.
Peabody Developmental Motor Scale | 12 weeks
  Peabody Developmental Motor Scales (PDMS-2) is composed of six subtests that measure interrelated abilities in early motor development. It was designed to assess gross and fine motor skills in children from birth through five years of age. This subtest measures aspects of a child's ability to automatically react to environmental events. Because reflexes typically become integrated by the time a child is 12 months old, this subtest is given only to children ages 2 weeks through 11 months. It measures a child's ability to sustain control of the body within its center of gravity and retain equilibrium

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Bashir, MS, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Keer I, Colla S, Van Leeuwen K, Vlaskamp C, Ceulemans E, Hoppenbrouwers K, Desoete A, Maes B. Exploring parental behavior and child interactive engagement: A study on children with a significant cognitive and motor developmental delay. Res Dev Disabil. 2017 May;64:131-142. doi: 10.1016/j.ridd.2017.04.002. Epub 2017 Apr 10. PMID 28407535